CLINICAL TRIAL: NCT06521827
Title: The Role of Short Course of Palliative Radiation in Metastatic Cancer Rectum
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehdaa Khaled Mahmoud, resident doctor at radiotherapy department at south Egypt cancer institute, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRTH in rectal cancer
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Cancer Rectum
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- short course radiotherapy (Experimental): patients with metastatic rectal cancer will receive short course of radiotherapy befor staring chemotherapy
  Interventions: Radiation: short course radiotherapy

INTERVENTIONS:
Radiation: short course radiotherapy — short course palliative radiotherapy

SUMMARY:
Short-course radiotherapy (SCRT), which allows the delivery of 25 Gy in five daily fractions, has emerged as an attractive strategy for rectal cancer treatment. Surgery can safely be deferred after SCRT, allowing an opportunity to deliver chemotherapy (ChT) preoperatively rather than postoperatively. In cases of metastatic disease, this represents an effective treatment option to improve local control and avoid colostomy in a subset of patients.

DETAILED DESCRIPTION:
All patients will be under go complete history and physical examination, proctoscopy and biopsy, followed by metastatic work up include chest X ray, pelvic abdominal CT.

Radiotherapy:

Target volume: all the gross primary disease and gross nodal involved plus 2 cm safety margin will be included. not involved node will not be included.

Dosage: total dose of 25 Gy over 5 fractions through 1 weak will be given. Time: Radiotherapy will be given first and chemotherapy will be given after 1 weak rest to avoid the over lapping toxicity.

Chemo therapy:

To be started after 1 weak rest after radiotherapy. CAPOX (oxaliplatin given intravenously at 130 mg/m2 on day 1, followed by oral capecitabine 1000 mg/m2 twice daily on days 1-14, in a 3-week cycle). or folfox (leucovorin calcium (IV 200 mg/m2 on day 1,2,15,16 ) + 5 fluorouracil (IV 600 mg/m2 on day 1,2,15,16)+ oxaliplatin (IV 85 mg/m2 on day 1, 15) plus target agent according to RAS status if wild for bevacizumab ( IV 5 ml/kg on day 1, 15) or cetiximab (IV 250 mg/m2 on day 1,8,15, 22) or vectibex (IV 6mg/kg on day 1,15)

Surgery:

Surgery if complete bowel obstruction as palliation or as treatment if controlled metastatic sites and primary

Follow up:

CT pelvi-abdomen will be done after 3 cycle of chemotherapy to assess the response then after end of CTH every 3 month in first year. Toxicity of RTH will be collected before and after RTH.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma pathological evidence in rectal carcinoma.
2. Metastatic unresectable rectal cancer.
3. Symptomatic disease for at least one of the following signs: bleeding, pain, tenesmus, obstruction,

Exclusion Criteria:

1. Previous radiotherapy.
2. Concomitant chemotherapy.
3. Previously created stoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The role of short course of palliative radiation in metastatic cancer rectum. | one year
  The role of short course of palliative radiation in metastatic cancer rectum.

REFERENCES:
- [Background] Santucci C, Mignozzi S, Malvezzi M, Boffetta P, Collatuzzo G, Levi F, La Vecchia C, Negri E. European cancer mortality predictions for the year 2024 with focus on colorectal cancer. Ann Oncol. 2024 Mar;35(3):308-316. doi: 10.1016/j.annonc.2023.12.003. Epub 2024 Jan 28. PMID 38286716
- [Background] Flyum IR, Mahic S, Grov EK, Joranger P. Health-related quality of life in patients with colorectal cancer in the palliative phase: a systematic review and meta-analysis. BMC Palliat Care. 2021 Sep 16;20(1):144. doi: 10.1186/s12904-021-00837-9. PMID 34530833
- [Background] Yoo RN, Cho HM, Kye BH. Management of obstructive colon cancer: Current status, obstacles, and future directions. World J Gastrointest Oncol. 2021 Dec 15;13(12):1850-1862. doi: 10.4251/wjgo.v13.i12.1850. PMID 35070029
- [Background] van Hooft JE, Veld JV, Arnold D, Beets-Tan RGH, Everett S, Gotz M, van Halsema EE, Hill J, Manes G, Meisner S, Rodrigues-Pinto E, Sabbagh C, Vandervoort J, Tanis PJ, Vanbiervliet G, Arezzo A. Self-expandable metal stents for obstructing colonic and extracolonic cancer: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2020. Endoscopy. 2020 May;52(5):389-407. doi: 10.1055/a-1140-3017. Epub 2020 Apr 7. PMID 32259849
- [Background] Tissera NS, Freile B, Waisberg F, Esteso F, Galli M, Loria FS, Luca R, Pedraza II, Enrico DH, Chacon C, Huertas E, Chacon MR, O'Connor JM. Short-course radiotherapy for rectal cancer: real-world evidence in Argentina. Ecancermedicalscience. 2023 Jun 1;17:1555. doi: 10.3332/ecancer.2023.1555. eCollection 2023. PMID 37396101